CLINICAL TRIAL: NCT01756937
Title: A Six-month, Multi Center, Randomizied, Double Blind, Parallel-group,Placebo Controlled Study to Evaluate Efficacy and Safety of Imotun Capsule in Osteoarthritis of the Knee
Brief Title: Efficacy and Safety of Imotun Capsule in Osteoarthritis of the Knee
Acronym: ABSOLUTE-R
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 238KOA12G
Record Dates: First submitted 2012-10-30; First posted 2012-12-28 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis of the knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imotun (Active Comparator): 300.03mg/cap,orally, 1 capsule once daily for 24 weeks
  Interventions: Drug: Imotun
- Placebo (Placebo Comparator): 1 capsule once daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Imotun — 300.03mg/cap,orally, 1 capsule once daily for 24 weeks
  Other Names: Avocado-Soya Unsaponifiables 300.03mg/Cap
  Arms: Imotun
Drug: Placebo — 1 capsule once daily for 24 weeks
  Arms: Placebo

SUMMARY:
Efficacy and safety of Imotun capsule in osteoarthritis of the knee

DETAILED DESCRIPTION:
A six-month, multi center, randomizied, double blind, parallel-group,placebo controlled study to evaluate efficacy and safety of Imotun capsule in osteoarthritis of the knee

ELIGIBILITY:
Inclusion Criteria:

* Agreement with written informed consent and 40 years of age and older
* Patients with more than 63months history of OA of knee according to ACR criteria
* Radiographic evidence of Kellgren & Lawrence grade II to III OA of the knee
* The 100mm Pain VAS is over 40mm
* The Lequensne's index is over 5

Exclusion Criteria:

* Treatment with SYSADOA within 3 months
* History of joint surgery within 5 years or Arthroscopic surgery within 1year
* Intra-articular injections within 3 months
* Treatment with NASIDs within 7 days
* Any history of adverse reaction to the study drugs
* clinically significant hepatic, renal, cardiovascular diseases
* Patients with gastrointestinal ulcers or bleeding disorders
* Pregnant women, nursing mothers or Fertile women who not practice contraception with appropriate methods
* History of drug abuse or alcoholism
* Patients on any other clinical trial or experimental treatment in the past 4 weeks
* An impossible one who participates in clinical trial by investigator's decision

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2013-01; Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Lequesne's index score at 24weeks | baseline, 24 weeks
  Change from baseline in the Lequesne's index score at 24weekS
100mm Pain VAS | 24 weeks
  assessment of 100mm Pain VAS (24weekS)

SECONDARY OUTCOMES:
Change from baseline Lequesne's index score at 4weeks | baseline, 4 weeks
  Change from baseline Lequesne's index score at 4weeks
Change from baseline Lequesne's index score at 8weeks | baseline, 8 weeks
  Change from baseline Lequesne's index score at 8weeks
Change from baseline Lequesne's index score at 16weeks | baseline, 16 weeks
  Change from baseline Lequesne's index score at 16weeks
100mm Pain VAS | 4weeks
  - Patient's assessment of 100mm Pain VAS
Global assement (Patient, Physician) | 4weeks
  -Global assement (Patient, Physician)
administration days of the rescue medication | 24weeks
  administration days of the rescue medication
The rate of patients who consumed the rescue medication | 24weeks
  The rate of patients who consumed the rescue medication
100mm Pain VAS | 8weeks
  - Patient's assessment of 100mm Pain VAS
100mm Pain VAS | 16weeks
  - Patient's assessment of 100mm Pain VAS
change from baseline 100mm Pain VAS at 4weeeks | baseline, 4weeks
  change from baseline 100mm Pain VAS at 4weeeks
change from baseline 100mm Pain VAS at 8weeeks | baseline, 8weeks
  change from baseline 100mm Pain VAS at 8weeeks
change from baseline 100mm Pain VAS at 16weeeks | baseline, 16 weeks
  change from baseline 100mm Pain VAS at 16weeeks
change from baseline 100mm Pain VAS at 24weeeks | baseline, 24 weeks
  change from baseline 100mm Pain VAS at 24weeeks
Global assement (Patient, Physician) | 8weeks
  -Global assement (Patient, Physician)
Global assement (Patient, Physician) | 16weeks
  -Global assement (Patient, Physician)
change from baseline Global assement (Patient, Physician) | baseline, 16weeks
  -Global assement (Patient, Physician)
Global assement (Patient, Physician) | 24weeks
  -Global assement (Patient, Physician)
dosing quantity of the rescue medication | 24weeks
  dosing quantity of the rescue medication

OTHER OUTCOMES:
Safety assessed by the incidence of adverse event | up to 24weeks
  Safety assessed by the incidence of adverse event
laboratory test | up to 24weeks
  laboratory test
medication history | up to 24weeks
  medication history

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyun Yoo, Principal Investigator — Hanyang University
Locations (9):
- South Korea (9):
  - Hallym Universicy Sacred heart Hospital, Anyang
  - Dong-A university Hospital, Busan
  - Yeungnam university medical center, Daegu
  - Chungnam National University hospital, Daejeon
  - Chonnam National university medical school & Hospital, Gwangju
  - hanyang University Guri Hospital, Gyeonggi-do
  - Konkuk University Medical Center, Seoul
  - Chung-Ang University hospital, Seoul
  - Hanyang University Hospital, Special City of Seoul